CLINICAL TRIAL: NCT00729937
Title: Strategies Using Off-Patent Antibiotics for Methicillin-Resistant Staphylococcus Aureus ("STOP MRSA") - A Phase IIB, Multi-Center, Randomized, Double-Blind Clinical Trial
Brief Title: Strategies Using Off-Patent Antibiotics for Methicillin Resistant S. Aureus "STOP MRSA"
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-0040
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Results first posted 2014-05-28 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2013-09

CONDITIONS: Staphylococcal Infection
Keywords: Methicillin, Staphylococcus aureus, MRSA
MeSH Terms: conditions — Staphylococcal Infections | interventions — Cephalexin; Clindamycin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- TMP/SMX vs. Placebo (Experimental): Subjects with an acute uncomplicated cutaneous abscess will be randomized to receive either Trimethoprim/Sulfamethoxazole (TMP/SMX) (4 single strength pills, 80 mg/400 mg each, twice per day) or 4 placebo pills (twice per day).
  Interventions: Other: Placebo; Drug: Trimethoprim-sulfamethoxazole
- TMP/SMX vs. Clindamycin (Experimental): Subjects with an acute uncomplicated wound infection will be randomized to receive Trimethoprim/Sulfamethoxazole (TMP/SMX) (4 single strength pills, 80 mg/400 mg each, twice per day, with alternating 1 identical placebo pill, twice per day) or clindamycin (300 mg, four times per day, with 3 placebo pills on alternating doses).
  Interventions: Drug: Clindamycin; Other: Placebo; Drug: Trimethoprim-sulfamethoxazole
- Cephalexin and TMP/SMX vs. Cephalexin (Experimental): Subjects with acute uncomplicated cellulitis will be randomized to receive cephalexin (500 mg, four times per day) and Trimethoprim/Sulfamethoxazole (TMP/SMX) (4 single strength pills, 80 mg/400 mg each, twice per day) or cephalexin (500 mg, four times per day) and placebo (4 pills, twice per day).
  Interventions: Drug: Cephalexin; Other: Placebo; Drug: Trimethoprim-sulfamethoxazole

INTERVENTIONS:
Drug: Cephalexin — 500 mg, four times per day.
  Arms: Cephalexin and TMP/SMX vs. Cephalexin
Drug: Clindamycin — 300 mg, four times per day.
  Arms: TMP/SMX vs. Clindamycin
Other: Placebo — Placebo tablet administered orally.
Drug: Trimethoprim-sulfamethoxazole — 4 single strength Trimethoprim/Sulfamethoxazole (TMP/SMX), 80 mg/400 mg each, twice per day.

SUMMARY:
The purpose of this study is to determine the optimal outpatient treatment strategy of uncomplicated skin and soft tissue infection (SSTI) in areas of the United States where the prevalence of Community-Acquired Methicillin-Resistant Staphylococcus (S.) aureus (CA-MRSA) is high. Infection with the S. aureus bacteria that is resistant to antibiotics is a cause of SSTIs. Three oral antibiotics will be tested for off patent treatment. Patients will receive Trimethoprim/Sulfamethoxazole (TMP/SMX), placebo (substance containing no medication), clindamycin, or cephalexin or some combination of these. The study population will include 2,235 volunteers, children 13 years of age and over and adults presenting to 5 large urban Emergency Departments. Therapy for acute uncomplicated SSTIs, including abscess, infected wound, and cellulitis will start on the day of enrollment. Participants may be involved in study related procedures for about 9 weeks.

DETAILED DESCRIPTION:
Community-acquired methicillin-resistant Staphylococcus aureus (CA-MRSA) has recently emerged as a cause of skin and soft-tissue infection (SSTI). In the current era of increasing CA-MRSA infections, the outpatient management of SSTIs has not been well studied. This will be a clinical trial to evaluate oral off-patent antibiotics for outpatient treatment of patients with any of the 3 main types of acute uncomplicated SSTI, i.e., abscesses, infected wounds, and cellulitis. Upon enrollment, subjects will be stratified by type of infection, and then randomized to various treatments. Subjects with an acute uncomplicated cutaneous abscess receiving incision and drainage (I&D) will be treated with Trimethoprim/Sulfamethoxazole (TMP/SMX) or placebo to determine whether the addition of an antibiotic with activity against CA-MRSA is more clinically efficacious than I&D alone. Subjects with an acute wound infection will be treated with TMP/SMX or clindamycin to determine if clindamycin, an antibiotic with activity against CA-MRSA, methicillin-susceptible Staphylococcus aureus (MSSA), and streptococci is more clinically efficacious than TMP/SMX, an antibiotic with activity against CA-MRSA and MSSA. Subjects with acute cellulitis will be treated with cephalexin/TMP/SMX or cephalexin/placebo to determine if cephalexin/TMP/SMX is more clinically efficacious than cephalexin alone. The primary objectives for each type of SSTI studied are to compare the cure rates in the per protocol (PP) population. Secondary objectives provide additional means of assessment for the clinical efficacy of the employed interventions and resolution of the infection and include describing microbiological cure, change in the dimension of erythema, composite cure, surgical procedures, invasive and recurrent infections, infections in household contacts, and time to normal activity and until analgesics are no longer used at various times in the PP/ modified intent-to-treat (mITT) populations. This is a multi-center, randomized, double-blind clinical trial in which subjects will be stratified by the type of infection and then randomized to various 7-day oral antibiotic treatments, including placebo-controlled and comparative designs. The study population will include children 13 years of age and over and adults, who weigh greater than or equal to 40 kg presenting to 5 large urban emergency departments. Therapy will start on the day of enrollment. Subjects will be evaluated upon enrollment, at 2-3 days after enrollment (OTV), at 1-3 days after the end-of-therapy (EOT), at 7-14 days after the end-of-therapy (TOC), and at 6-8 weeks after the end-of-therapy (EFV).

ELIGIBILITY:
Inclusion Criteria:

* Adult or child 13 years of age and older (who weighs greater than or equal to 40 kg);
* Have a skin and soft tissue infection (SSTI) with all three local findings of erythema (> 2 cm across the lesion or from a discrete wound edge), tenderness, and swelling/induration. Fever, leukocytosis, and lymphangitis will be noted, but are not enrollment criteria. SSTI with these local findings will be further categorized and defined as one of:

  1. Abscess - a fluctuant and/or indurated lesion, or findings of a fluid-filled cavity on soft tissue ultrasound evaluation that, when opened reveals purulent material, receiving incision and drainage (I&D) (considered standard care for abscess) and having a minimum diameter (along any axis) of at least 2 cm (measured from the borders of induration, if a fluctuant lesion, or borders of the abscess cavity on ultrasound, if not fluctuant).

     Note: Although I&D of an abscess is considered standard care (i.e., patients will receive I&D whether or not they are enrolled in the study), the procedure may be performed after enrollment into the study so that prior measurements of the area of erythema and swelling/induration can be obtained unless it is an occult abscess in which the I&D will be performed prior to enrollment to verify infection type and ensure correct classification of the subject.
  2. Infected Wound - a wound (defined as any apparent break in the skin) with any apparent drainage limited in depth to only involving skin and subcutaneous tissue, including sutured cutaneous wounds not involving intra-abdominal surgeries contaminated with bacterial or bowel contents (e.g., colon surgery and empyema drainage), and
  3. Cellulitis - an area of erythema without the presence of a wound with drainage or abscess; Cellulitis associated with an abscess will be categorized as an abscess. Cellulitis associated with an infected wound will be classified as an infected wound. Patients with cellulitis and an abscess less than 2 cm will be excluded. Infected wound associated with an abscess that may require I&D, will be classified as an infected wound.
* Have the infected lesion for 7 days or less duration;
* Are to receive outpatient treatment at enrollment/baseline;
* Express willingness and ability to be contacted and return for re-evaluation according to the study protocol;
* Provide written informed consent (and for subjects ages 13-17, consent from their guardian and assent);
* Negative pregnancy test for subjects who are women of childbearing potential.

Exclusion Criteria:

* Severe allergy or reaction to study drug or drugs similar to the study drug relevant to whichever study sub-trial the subject would be assigned to (e.g., patients with severe or life-threatening penicillin allergies, allergy to any cephalosporin, clindamycin, or sulfonamides, or any other drug containing sulfur such as thiazides, furosemide, and oral sulfonylureas);
* Concomitant treatment (i.e., while on study drug therapy) with coumadin, phenytoin, or methotrexate, or suspected G-6-PD or folic acid deficiency;
* Expected inability to swallow or absorb the study drug (assessed by patient history);
* Pregnancy, nursing, or expectation of becoming pregnant while on study drug;
* Perirectal (within 5 cm of anus), perineal non-skin lesions (i.e., mucosal), or paronychial location of infection. Scrotal and labial abscesses will not be excluded.
* An infection due to a mammalian bite;
* Treatment with a study drug relevant to their infection type, or another systemic antibiotic in the previous 48 hours (i.e., before screening/baseline) unless associated with treatment failure which is defined as a patient who has been on prior (non study drug) antibiotics for at least 72 hours and failed.
* Expected concurrent treatment with a topical antibiotic or another systemic antibiotic up to Test-of-Cure Visit (TOC) (note: if patient was using a topical antibiotic previously, they can still be enrolled if they agree to stop using it);
* Immunodeficiency [e.g., absolute neutrophil count <500/mm^3, chronic immunosuppressive drugs, active chemotherapy, or known acquired immunodeficiency syndrome (AIDS) (CD4 count <200 or AIDS-defining illness within the last year) assessed by patient history]. Note: patients who had prior AIDS-defining illness or CD4 count <200 in the past may be enrolled if most recent CD4 count >200;
* Burn or active chronic skin condition (e.g., including rash or eczema) related to the skin and soft-tissue infection (SSTI) at screening/baseline;
* Infection related to currently indwelling device (e.g., intravenous line), excepting sutures associated with qualifying infected wounds which will be removed upon enrollment;
* Infection for which prior cultures reveal in vitro resistance of a pathogen to a study drug in the previous month prior to screening/baseline;
* Known or suspected osteomyelitis or septic arthritis;
* Infection related to diabetic foot, decubitus, or ischemic ulcer;
* Known severe renal insufficiency (creatinine clearance < 50 mL/min) calculated by measurement of serum creatinine if patient provides this history or based on past studies at baseline/enrollment;
* Prior enrollment in this study within 12 weeks;
* Another active infection of another organ system (e.g., pneumonia) or more than one active (i.e., currently on antibiotic treatment and/or requiring I&D) SSTI site (e.g., a site noncontiguous with the infection under study). Note: Minor folliculitis at secondary site is not an exclusion;
* Presence of an abscess that has completely drained, either spontaneously or by a healthcare provider prior to enrollment;
* An infected wound or cellulitis that has been surgically explored (>1 cm incision) and does not reveal an abscess. Cellulitis that has been needled, minimally incised (less than or equal to 1 cm) or punch biopsied and no purulent drainage found can still be enrolled;
* Currently incarcerated in a detention facility or in police custody (note: patients wearing a monitoring device can be enrolled) at baseline/screening;
* For patients with an infected wound, history of C. difficile infection, pseudomembranous colitis, or active diarrhea at baseline/screening;
* For patients with an infected wound, severe liver disease based on patient history;
* An intravenous (IV) drug user in the last month with current presence of fever;
* Current residence in a nursing home or other long term care facility at baseline/screening;
* Expected use of other investigational drug or vaccine while on study drug;
* For patients with an abscess, cardiac conditions associated with the highest risk of adverse outcome from endocarditis for which prophylaxis is reasonable, including patients with prosthetic cardiac valve or prosthetic material used for cardiac valve repair, history of previous infective endocarditis, congenital heart disease (excluding mitral valve prolapse), and history of cardiac transplantation recipients who develop cardiac valvulopathy;
* Presence of an organic foreign body, e.g., wood (note: subjects with embedded non-organic materials, e.g., metal or glass, that can be completely removed can still be enrolled if physician is certain there is no foreign body left).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2265 (Actual)
Dates: Start 2009-04; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Maricopa Medical Center - Emergency Medicine, Phoenix, Arizona
  - University of California Los Angeles - Olive View Medical Center, Sylmar, California
  - Johns Hopkins University at Mount Washington - Emergency Medicine, Baltimore, Maryland
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Temple University Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Mower WR, Crisp JG, Krishnadasan A, Moran GJ, Abrahamian FM, Lovecchio F, Karras DJ, Steele MT, Rothman RE, Talan DA. Effect of Initial Bedside Ultrasonography on Emergency Department Skin and Soft Tissue Infection Management. Ann Emerg Med. 2019 Sep;74(3):372-380. doi: 10.1016/j.annemergmed.2019.02.002. Epub 2019 Mar 27. PMID 30926187
- [Derived] Talan DA, Moran GJ, Krishnadasan A, Abrahamian FM, Lovecchio F, Karras DJ, Steele MT, Rothman RE, Mower WR. Subgroup Analysis of Antibiotic Treatment for Skin Abscesses. Ann Emerg Med. 2018 Jan;71(1):21-30. doi: 10.1016/j.annemergmed.2017.07.483. Epub 2017 Oct 5. PMID 28987525
- [Derived] Moran GJ, Krishnadasan A, Mower WR, Abrahamian FM, LoVecchio F, Steele MT, Rothman RE, Karras DJ, Hoagland R, Pettibone S, Talan DA. Effect of Cephalexin Plus Trimethoprim-Sulfamethoxazole vs Cephalexin Alone on Clinical Cure of Uncomplicated Cellulitis: A Randomized Clinical Trial. JAMA. 2017 May 23;317(20):2088-2096. doi: 10.1001/jama.2017.5653. PMID 28535235
- [Derived] Talan DA, Lovecchio F, Abrahamian FM, Karras DJ, Steele MT, Rothman RE, Krishnadasan A, Mower WR, Hoagland R, Moran GJ. A Randomized Trial of Clindamycin Versus Trimethoprim-sulfamethoxazole for Uncomplicated Wound Infection. Clin Infect Dis. 2016 Jun 15;62(12):1505-1513. doi: 10.1093/cid/ciw177. Epub 2016 Mar 29. PMID 27025829
- [Derived] Talan DA, Mower WR, Krishnadasan A, Abrahamian FM, Lovecchio F, Karras DJ, Steele MT, Rothman RE, Hoagland R, Moran GJ. Trimethoprim-Sulfamethoxazole versus Placebo for Uncomplicated Skin Abscess. N Engl J Med. 2016 Mar 3;374(9):823-32. doi: 10.1056/NEJMoa1507476. PMID 26962903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between 13APR2009 and 16APR2013 from those who presented with an abscess, infected wound, or cellulitis at emergency departments at each of the clinical sites.
Groups:
- Abscess, Placebo: Participants with an acute uncomplicated cutaneous abscess received 4 placebo pills twice per day.
- Abscess, TMP/SMX: Participants with an acute uncomplicated cutaneous abscess received Trimethoprim/Sulfamethoxazole (TMP/SMX) as 4 single strength pills of 80mg/400mg each, twice per day.
- Infected Wound, TMP/SMX: Participants with an acute uncomplicated wound infection received Trimethoprim/Sulfamethoxazole (TMP/SMX) as 4 single strength pills of 80mg/400mg each, twice per day, with alternating 1 identical placebo pill, twice per day.
- Infected Wound, Clindamycin: Participants with an acute uncomplicated wound infection received clindamycin as 300 mg pills, four times per day, with 3 placebo pills on alternating doses.
- Cellulitis, Cephalexin and TMP/SMX: Participants with acute uncomplicated cellulitis received cephalexin as 500 mg pills, four times per day, and Trimethoprim/Sulfamethoxazole (TMP/SMX) as 4 single strength pills of 80mg/400mg each, twice per day.
- Cellulitis, Cephalexin: Participants with acute uncomplicated cellulitis received cephalexin as 500 mg pills, four times per day, and 4 placebo pills, twice per day.
Period: Overall Study
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Started | 629 | 636 | 251 | 249 | 249 | 251
Completed | 555 | 548 | 222 | 215 | 221 | 214
Not Completed | 74 | 88 | 29 | 34 | 28 | 37
Not completed — Lost to Follow-up | 49 | 58 | 18 | 33 | 18 | 23
Not completed — Physician Decision | 7 | 16 | 2 | 0 | 5 | 8
Not completed — Death | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 5 | 6 | 0 | 4 | 2
Not completed — Randomized but not treated | 12 | 6 | 1 | 0 | 1 | 3
Not completed — Did not meet eligibility criteria | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Incarcerated | 0 | 2 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is the per protocol population. All participants who met enrollment criteria, had none of the exclusion criteria, completed at least 75% of the first 5 days of antimicrobial therapy, and had physical follow-up at the Test of Cure (TOC) visit were included in the per protocol population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin | Total
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193 | 1869
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (12.3) | 37.0 (12.6) | 40.4 (13.1) | 38.0 (13.3) | 39.7 (13.3) | 39.4 (13.2) | 38.0 (12.9)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 10 | 3 | 5 | 3 | 2 | 40
  Between 18 and 65 years | 513 | 511 | 191 | 195 | 206 | 187 | 1803
  >=65 years | 3 | 3 | 4 | 3 | 9 | 4 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 225 | 221 | 65 | 81 | 81 | 90 | 763
  Male | 308 | 303 | 133 | 122 | 137 | 103 | 1106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 0 | 2 | 2 | 0 | 9
  Asian | 2 | 5 | 0 | 0 | 2 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 233 | 232 | 71 | 73 | 75 | 68 | 752
  White | 252 | 244 | 115 | 117 | 123 | 111 | 962
  More than one race | 22 | 22 | 7 | 3 | 7 | 8 | 69
  Unknown or Not Reported | 21 | 18 | 5 | 8 | 9 | 4 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 180 | 178 | 63 | 72 | 75 | 60 | 628
  Not Hispanic or Latino | 353 | 346 | 134 | 131 | 143 | 133 | 1240
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 533 | 524 | 198 | 203 | 218 | 193 | 1869

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Clinical Cure as of the TOC Visit in the Intent to Treat Population
Description: Clinical cure at TOC was defined as no failure on any previous visit up through the TOC, absence of fever, and resolution or minimal presence of all the following signs and symptoms from baseline based on clinician assessment of erythema, swelling, and tenderness. A participant would have been a clinical failure at the On Therapy (OTV) visit with presence of fever attributable to the infection being studied, increase in erythema by 25% or more, or worsening of both swelling and tenderness based on clinical assessment. A participant would have been a clinical failure at the End of Therapy (EOT) visit with presence of fever attributable to the infection being studied, increase or no improvement in erythema, or no improvement in either swelling or tenderness based on clinical assessment.
Time Frame: Days 14-21
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 617 | 630 | 250 | 249 | 248 | 248
participants
  Clinical Cure | 454 | 507 | 197 | 198 | 189 | 171
  Clinical Failure | 163 | 123 | 53 | 51 | 59 | 77

2. Primary Outcome: Number of Participants With Clinical Cure as of the Test-of-Cure (TOC) Visit in the Per Protocol Population
Description: as for outcome 1
Time Frame: Days 14-21
Population: The analysis population is the per protocol population. All participants who met enrollment criteria, had none of the exclusion criteria, completed at least 75% of the first 5 days of antimicrobial therapy, and had physical follow-up at the Test of Cure (TOC) visit were included in the per protocol population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193
participants
  Clinical Cure | 457 | 487 | 182 | 187 | 182 | 165
  Clinical Failure | 76 | 37 | 16 | 16 | 36 | 28

3. Secondary Outcome: Number of Participants With Reduction in Erythema Dimensions by 5% Intervals at the On-therapy Visit in the Per Protocol Population
Description: The area of erythema was measured in square centimeters at baseline and at the on-therapy visit. For each subject, the change in area was calculated as the area at on-therapy subtracted from the area at baseline. The change in area was then divided by the original area to determine the proportional change. Participants were then categorized by reductions in 5% intervals, with participants whose erythema did not change or increased categorized as no reduction.
Time Frame: Day 1 to Day 3-4
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 523 | 195 | 203 | 217 | 192
participants
  No reduction | 59 | 37 | 11 | 17 | 30 | 33
  >0%-5% reduction | 3 | 2 | 1 | 1 | 1 | 2
  >5%-10% reduction | 1 | 4 | 3 | 0 | 5 | 1
  >10%-15% reduction | 3 | 3 | 1 | 3 | 5 | 0
  >15%-20% reduction | 2 | 6 | 4 | 5 | 3 | 2
  >20%-25% reduction | 6 | 3 | 5 | 2 | 4 | 4
  >25%-30% reduction | 11 | 6 | 5 | 3 | 5 | 3
  >30%-35% reduction | 13 | 7 | 4 | 5 | 2 | 7
  >35%-40% reduction | 12 | 13 | 3 | 3 | 6 | 2
  >40%-45% reduction | 16 | 15 | 7 | 6 | 8 | 6
  >45%-50% reduction | 12 | 12 | 5 | 6 | 5 | 9
  >50%-55% reduction | 13 | 6 | 6 | 6 | 4 | 6
  >55%-60% reduction | 10 | 10 | 4 | 2 | 9 | 8
  >60%-65% reduction | 14 | 21 | 12 | 6 | 15 | 3
  >65%-70% reduction | 19 | 9 | 6 | 5 | 7 | 7
  >70%-75% reduction | 14 | 17 | 8 | 7 | 9 | 5
  >75%-80% reduction | 13 | 21 | 6 | 16 | 8 | 7
  >80%-85% reduction | 19 | 18 | 8 | 3 | 10 | 6
  >85%-90% reduction | 18 | 13 | 4 | 8 | 5 | 8
  >90%-95% reduction | 13 | 16 | 5 | 10 | 5 | 6
  >95%-100% reduction | 262 | 284 | 87 | 89 | 71 | 67

4. Secondary Outcome: Number of Participants With Reduction in Erythema Dimensions by 5% Intervals at the On-therapy Visit in the Intent to Treat Population
Description: as for outcome 3
Time Frame: Day 1 to Day 3-4
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 604 | 599 | 237 | 241 | 237 | 230
participants
  No reduction | 67 | 43 | 12 | 18 | 34 | 41
  >0%-5% reduction | 3 | 2 | 1 | 1 | 1 | 2
  >5%-10% reduction | 2 | 4 | 3 | 1 | 6 | 1
  >10%-15% reduction | 3 | 3 | 1 | 4 | 5 | 0
  >15%-20% reduction | 2 | 7 | 4 | 5 | 5 | 2
  >20%-25% reduction | 7 | 5 | 6 | 3 | 4 | 5
  >25%-30% reduction | 12 | 6 | 5 | 4 | 5 | 3
  >30%-35% reduction | 13 | 8 | 5 | 6 | 4 | 7
  >35%-40% reduction | 12 | 15 | 3 | 4 | 6 | 6
  >40%-45% reduction | 20 | 17 | 8 | 7 | 9 | 6
  >45%-50% reduction | 13 | 15 | 6 | 6 | 5 | 10
  >50%-55% reduction | 14 | 7 | 7 | 8 | 4 | 9
  >55%-60% reduction | 12 | 11 | 4 | 2 | 9 | 8
  >60%-65% reduction | 15 | 24 | 12 | 7 | 16 | 4
  >65%-70% reduction | 21 | 10 | 7 | 6 | 7 | 9
  >70%-75% reduction | 18 | 20 | 10 | 9 | 11 | 6
  >75%-80% reduction | 17 | 22 | 11 | 17 | 9 | 8
  >80%-85% reduction | 20 | 20 | 9 | 3 | 11 | 6
  >85%-90% reduction | 20 | 16 | 5 | 11 | 6 | 9
  >90%-95% reduction | 15 | 16 | 7 | 11 | 6 | 8
  >95%-100% reduction | 298 | 328 | 111 | 108 | 74 | 80

5. Secondary Outcome: Number of Participants With Reduction in Erythema Dimensions by 5% Intervals at the End-of-therapy Visit in the Per Protocol Population
Description: The area of erythema was measured in square centimeters at baseline and at the end-of-therapy visit. For each subject, the change in area was calculated as the area at end-of-therapy subtracted from the area at baseline. The change in area was then divided by the original area to determine the proportional change. Participants were then categorized by reductions in 5% intervals, with participants whose erythema did not change or increased categorized as no reduction.
Time Frame: Day 1 to Day 8-10
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 527 | 520 | 193 | 200 | 212 | 190
participants
  No reduction | 4 | 3 | 3 | 3 | 5 | 5
  >0%-5% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >5%-10% reduction | 1 | 0 | 0 | 0 | 1 | 0
  >10%-15% reduction | 0 | 1 | 1 | 0 | 0 | 0
  >15%-20% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >20%-25% reduction | 0 | 0 | 0 | 0 | 1 | 0
  >25%-30% reduction | 2 | 1 | 1 | 0 | 0 | 1
  >30%-35% reduction | 0 | 1 | 0 | 0 | 1 | 1
  >35%-40% reduction | 2 | 1 | 0 | 0 | 1 | 0
  >40%-45% reduction | 0 | 3 | 2 | 0 | 0 | 1
  >45%-50% reduction | 2 | 0 | 1 | 1 | 0 | 0
  >50%-55% reduction | 4 | 1 | 2 | 1 | 0 | 2
  >55%-60% reduction | 0 | 5 | 1 | 1 | 1 | 2
  >60%-65% reduction | 1 | 0 | 3 | 2 | 5 | 1
  >65%-70% reduction | 4 | 3 | 2 | 1 | 2 | 2
  >70%-75% reduction | 3 | 2 | 3 | 0 | 5 | 2
  >75%-80% reduction | 6 | 2 | 2 | 1 | 2 | 2
  >80%-85% reduction | 4 | 5 | 1 | 3 | 0 | 1
  >85%-90% reduction | 7 | 7 | 1 | 4 | 4 | 4
  >90%-95% reduction | 9 | 7 | 3 | 1 | 1 | 4
  >95%-100% reduction | 478 | 478 | 167 | 182 | 183 | 162

6. Secondary Outcome: Number of Participants With Reduction in Erythema Dimensions by 5% Intervals at the End-of-therapy Visit in the Intent to Treat Population
Description: as for outcome 5
Time Frame: Day 1 to Day 8-10
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 582 | 576 | 228 | 231 | 229 | 225
participants
  No reduction | 5 | 3 | 3 | 3 | 5 | 5
  >0%-5% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >5%-10% reduction | 1 | 0 | 0 | 0 | 1 | 0
  >10%-15% reduction | 0 | 1 | 1 | 1 | 0 | 1
  >15%-20% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >20%-25% reduction | 0 | 0 | 1 | 0 | 1 | 0
  >25%-30% reduction | 2 | 1 | 1 | 0 | 0 | 1
  >30%-35% reduction | 0 | 1 | 0 | 0 | 1 | 1
  >35%-40% reduction | 2 | 1 | 0 | 0 | 1 | 0
  >40%-45% reduction | 0 | 3 | 3 | 0 | 0 | 1
  >45%-50% reduction | 2 | 0 | 1 | 1 | 0 | 0
  >50%-55% reduction | 4 | 1 | 2 | 1 | 0 | 2
  >55%-60% reduction | 0 | 5 | 1 | 1 | 1 | 2
  >60%-65% reduction | 2 | 0 | 3 | 2 | 5 | 2
  >65%-70% reduction | 4 | 3 | 2 | 1 | 2 | 3
  >70%-75% reduction | 3 | 2 | 3 | 2 | 5 | 2
  >75%-80% reduction | 6 | 2 | 2 | 1 | 3 | 2
  >80%-85% reduction | 4 | 5 | 1 | 4 | 0 | 2
  >85%-90% reduction | 7 | 9 | 2 | 4 | 4 | 6
  >90%-95% reduction | 9 | 7 | 5 | 2 | 2 | 7
  >95%-100% reduction | 531 | 532 | 197 | 208 | 198 | 188

7. Secondary Outcome: Number of Participants With Reduction in Erythema Dimensions by 5% Intervals at the TOC Visit in the Per Protocol Population
Description: The area of erythema was measured in square centimeters at baseline and at the TOC visit. For each subject, the change in area was calculated as the area at TOC subtracted from the area at baseline. The change in area was then divided by the original area to determine the proportional change. Participants were then categorized by reductions in 5% intervals, with participants whose erythema did not change or increased categorized as no reduction.
Time Frame: Day 1 to Day 14-21
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 532 | 521 | 197 | 201 | 215 | 192
participants
  No reduction | 2 | 0 | 1 | 1 | 2 | 0
  >0%-5% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >5%-10% reduction | 0 | 0 | 0 | 0 | 0 | 1
  >10%-15% reduction | 0 | 0 | 1 | 0 | 0 | 0
  >15%-20% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >20%-25% reduction | 0 | 1 | 0 | 0 | 0 | 0
  >25%-30% reduction | 0 | 0 | 1 | 0 | 0 | 0
  >30%-35% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >35%-40% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >40%-45% reduction | 0 | 0 | 0 | 0 | 1 | 0
  >45%-50% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >50%-55% reduction | 0 | 0 | 1 | 0 | 0 | 0
  >55%-60% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >60%-65% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >65%-70% reduction | 0 | 0 | 1 | 0 | 1 | 0
  >70%-75% reduction | 0 | 0 | 1 | 0 | 2 | 1
  >75%-80% reduction | 2 | 0 | 0 | 0 | 1 | 1
  >80%-85% reduction | 0 | 2 | 0 | 0 | 1 | 0
  >85%-90% reduction | 4 | 1 | 0 | 0 | 0 | 0
  >90%-95% reduction | 4 | 1 | 0 | 1 | 0 | 0
  >95%-100% reduction | 520 | 516 | 191 | 199 | 207 | 189

8. Secondary Outcome: Number of Participants With Reduction in Erythema Dimensions by 5% Intervals at the TOC Visit in the Intent to Treat Population
Description: as for outcome 7
Time Frame: Day 1 to Day 14-21
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 573 | 565 | 223 | 223 | 228 | 221
participants
  No reduction | 2 | 0 | 1 | 1 | 2 | 0
  >0%-5% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >5%-10% reduction | 0 | 0 | 0 | 0 | 0 | 1
  >10%-15% reduction | 0 | 0 | 1 | 0 | 0 | 0
  >15%-20% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >20%-25% reduction | 0 | 1 | 0 | 0 | 0 | 0
  >25%-30% reduction | 0 | 0 | 1 | 1 | 0 | 0
  >30%-35% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >35%-40% reduction | 0 | 0 | 0 | 0 | 0 | 1
  >40%-45% reduction | 0 | 0 | 0 | 0 | 1 | 0
  >45%-50% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >50%-55% reduction | 0 | 0 | 1 | 0 | 0 | 0
  >55%-60% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >60%-65% reduction | 0 | 0 | 0 | 0 | 0 | 0
  >65%-70% reduction | 0 | 0 | 1 | 1 | 1 | 0
  >70%-75% reduction | 0 | 0 | 1 | 0 | 2 | 1
  >75%-80% reduction | 2 | 1 | 0 | 0 | 1 | 1
  >80%-85% reduction | 0 | 2 | 0 | 0 | 1 | 0
  >85%-90% reduction | 4 | 1 | 0 | 0 | 0 | 0
  >90%-95% reduction | 4 | 1 | 1 | 1 | 0 | 0
  >95%-100% reduction | 561 | 559 | 216 | 219 | 220 | 217

9. Secondary Outcome: Number of Participants by Composite Clinical Outcome at the TOC Visit in the Per Protocol Population
Description: Participants were categorized as composite clinical cure if they had resolution of all symptoms/signs of infection, or improvement to such an extent that no additional antibiotic therapy and/or surgical procedures were necessary. Participants were categorized as composite clinical failure if they had lack of resolution of all signs and symptoms of infection to such an extent that further antibiotic therapy and/or surgical procedures were necessary.
Time Frame: Day 14-21
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193
participants
  Composite Clinical Cure | 396 | 453 | 113 | 114 | 160 | 149
  Composite Clinical Failure | 137 | 71 | 85 | 89 | 58 | 44

10. Secondary Outcome: Number of Participants With Each Microbiological Outcome at the TOC Visit in the Per Protocol Population
Description: Participants were categorized for the microbiological outcome with Presumed eradication if they were not deemed a clinical failure through TOC. Those who were deemed a clinical failure through the TOC were classified as one of the following: Persistence=persistent growth of a pre-therapy pathogen; New infection=growth of a new pathogen and eradication of initial pathogen; Super-infection=growth of a new pathogen in addition to persistent growth of pre-therapy pathogen; Unclassified=no specimen for culture or growth of a pathogen in subsequent culture specimen of cellulitis participants, or for whom initial culture specimens were negative or were not obtained for infected wound and abscess participants; or Indeterminate=not meeting any one of the above microbiologic outcome criteria.
Time Frame: Day 14-21
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193
participants
  Presumed eradication | 457 | 487 | 182 | 187 | 182 | 165
  Persistence | 39 | 15 | 5 | 6 | 0 | 0
  New infection | 1 | 0 | 2 | 1 | 0 | 0
  Super-infection | 8 | 4 | 0 | 0 | 0 | 0
  Unclassified | 28 | 18 | 9 | 9 | 13 | 11
  Indeterminate | 0 | 0 | 0 | 0 | 23 | 17

11. Secondary Outcome: Number of Participants Requiring Surgical Intervention Through the TOC Visit in the Per Protocol Population
Description: All surgical procedures such as incision and drainage (I&D) and debridement that were related to the current infection under study or significant to the health of the subject, except for the initial I&D of an abscess for participants in the abscess or infected wound arms, were recorded. Participants who required a surgical intervention between the initial enrollment (excluding the initial I&D as applicable) and the test-of-cure visit are summarized.
Time Frame: Day 1 through Day 14-21
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193
participants | 46 | 18 | 13 | 6 | 26 | 17

12. Secondary Outcome: Number of Participants Requiring Surgical Intervention Through the TOC Visit in the Intent to Treat Population
Description: as for outcome 11
Time Frame: Day 1 through Day 14-21
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 617 | 630 | 250 | 249 | 248 | 248
participants | 52 | 25 | 16 | 9 | 26 | 28

13. Secondary Outcome: Number of Participants Requiring Surgical Intervention Through the Extended Follow-up Visit (EFV) in the Per Protocol Population
Description: All surgical procedures such as incision and drainage (I&D) and debridement that were related to the current infection under study or significant to the health of the subject, except for the initial I&D of an abscess for participants in the abscess or infected wound arms, were recorded. Participants who required a surgical intervention between the initial enrollment (excluding the initial I&D as applicable) and the extended follow-up visit are summarized.
Time Frame: Day 1 through Day 49-63
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193
participants | 69 | 42 | 17 | 8 | 33 | 20

14. Secondary Outcome: Number of Participants Requiring Surgical Intervention Through the Extended Follow-up Visit (EFV) in the Intent to Treat Population
Description: as for outcome 13
Time Frame: Day 1 through Day 49-63
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 617 | 630 | 250 | 249 | 248 | 248
participants | 76 | 52 | 20 | 12 | 33 | 31

15. Secondary Outcome: Number of Participants With Development of an Invasive Infection Through the TOC Visit in the Per Protocol Population
Description: Participants were evaluated for invasive infection, which included, but was not limited to, findings of severe sepsis/septic shock, endocarditis, pneumonia, necrotizing soft tissue, osteomyelitis, and bacteremia. A positive response to at least one finding was considered invasive infection for this outcome measure.
Time Frame: Day 1 through Day 14-21
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193
participants | 0 | 1 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Development of an Invasive Infection Through the TOC Visit in the Intent to Treat Population
Description: as for outcome 15
Time Frame: Day 1 through Day 14-21
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 617 | 630 | 250 | 249 | 248 | 248
participants | 1 | 1 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Development of an Invasive Infection Through the EFV Visit in the Per Protocol Population
Description: as for outcome 15
Time Frame: Day 1 through Day 49-63
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193
participants | 2 | 2 | 0 | 0 | 1 | 0

18. Secondary Outcome: Number of Participants With Development of an Invasive Infection Through the EFV Visit in the Intent to Treat Population
Description: as for outcome 15
Time Frame: Day 1 through Day 49-63
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 617 | 630 | 250 | 249 | 248 | 248
participants | 3 | 2 | 0 | 0 | 1 | 0

19. Secondary Outcome: Number of Participants Who Developed a Recurrent Infection at the Original Infection Site Through the TOC Visit in the Per Protocol Population
Description: Participants were evaluated for the development of a recurrent, or repeat, infection at the original infection site. Participants who were reported to have developed a recurrent infection though the test-of-cure visit are summarized.
Time Frame: Day 1 through Day 14-21
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193
participants | 16 | 11 | 13 | 3 | 30 | 22

20. Secondary Outcome: Number of Participants Who Developed a Recurrent Infection at the Original Infection Site Through the TOC Visit in the Intent to Treat Population
Description: as for outcome 19
Time Frame: Day 1 through Day 14-21
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 617 | 630 | 250 | 249 | 248 | 248
participants | 17 | 13 | 15 | 4 | 32 | 29

21. Secondary Outcome: Number of Participants Who Developed a Recurrent Infection at the Original Infection Site Through the EFV Visit in the Per Protocol Population
Description: Participants were evaluated for the development of a recurrent, or repeat, infection at the original infection site. Participants who were reported to have developed a recurrent infection though the extended follow-up visit are summarized.
Time Frame: Day 1 through Day 49-63
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193
participants | 23 | 26 | 14 | 4 | 33 | 24

22. Secondary Outcome: Number of Participants Who Developed a Recurrent Infection at the Original Infection Site Through the EFV Visit in the Intent to Treat Population
Description: as for outcome 21
Time Frame: Day 1 through Day 49-63
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 617 | 630 | 250 | 249 | 248 | 248
participants | 26 | 30 | 16 | 6 | 35 | 31

23. Secondary Outcome: Number of Participants With Infections in Household Contacts Through the TOC Visit in the Per Protocol Population
Description: At each follow-up visit, participants were asked about history of skin infections in household members (e.g., similar skin infection in a family member). This outcome measure relied solely on participant reporting. Participants who reported having a family member with a similar infection though the test-of-cure visit are summarized.
Time Frame: Day 1 through Day 14-21
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193
participants | 22 | 9 | 1 | 5 | 6 | 4

24. Secondary Outcome: Number of Participants With Infections in Household Contacts Through the TOC Visit in the Intent to Treat Population
Description: as for outcome 23
Time Frame: Day 1 through Day 14-21
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 617 | 630 | 250 | 249 | 248 | 248
participants | 22 | 12 | 1 | 6 | 7 | 4

25. Secondary Outcome: Number of Participants With Infections in Household Contacts Through the EFV Visit in the Per Protocol Population
Description: At each follow-up visit, participants were asked about history of skin infections in household members (e.g., similar skin infection in a family member). This outcome measure relied solely on participant reporting. Participants who reported having a family member with a similar infection though the extended follow-up visit are summarized.
Time Frame: Day 1 through Day 49-63
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193
participants | 33 | 20 | 6 | 9 | 10 | 5

26. Secondary Outcome: Number of Participants With Infections in Household Contacts Through the EFV Visit in the Intent to Treat Population
Description: as for outcome 25
Time Frame: Day 1 through Day 49-63
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 617 | 630 | 250 | 249 | 248 | 248
participants | 35 | 25 | 6 | 11 | 11 | 5

27. Secondary Outcome: Number of Participants With Adverse Events Considered Associated With the Study Product by MedDRA System Organ Class
Description: All adverse events were recorded through the test of cure visit; serious adverse events and new and recurrent skin infections were recorded though the extended follow-up visit. All AEs were assessed for association with the study product by a clinician and were considered associated with study product if the event was temporally related to the administration of the study product and no other etiology more likely explains the event. Associated adverse events are summarized by MedDRA System Organ Class.
Time Frame: Day 1 through Day 49-63
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 617 | 630 | 250 | 249 | 248 | 248
participants
  Cardiac disorders | 0 | 0 | 0 | 1 | 0 | 0
  Eye disorders | 3 | 1 | 0 | 0 | 0 | 0
  Gastrointestinal disorders | 164 | 198 | 82 | 93 | 87 | 73
  General disorders and administration site conditio | 6 | 11 | 3 | 1 | 2 | 2
  Infections and infestations | 5 | 4 | 1 | 1 | 1 | 1
  Injury, poisoning and procedural complications | 1 | 0 | 0 | 0 | 0 | 0
  Investigations | 1 | 0 | 1 | 0 | 0 | 0
  Metabolism and nutrition disorders | 7 | 11 | 2 | 4 | 3 | 0
  Musculoskeletal and connective tissue disorders | 3 | 3 | 0 | 0 | 0 | 0
  Nervous system disorders | 38 | 44 | 16 | 15 | 16 | 20
  Psychiatric disorders | 0 | 1 | 0 | 0 | 0 | 0
  Renal and urinary disorders | 2 | 0 | 1 | 0 | 1 | 0
  Reproductive system and breast disorders | 1 | 0 | 0 | 1 | 1 | 0
  Respiratory, thoracic and mediastinal disorders | 3 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders | 10 | 14 | 5 | 6 | 15 | 7
  Vascular disorders | 2 | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Mean Days Missed From Normal Activities in the Per Protocol Population
Description: As a quality of life measure, participants maintained a memory aid from Day 1 to Day 14 to track measures such as participation in normal life activities. The maximum number of days assessed, 14, was assigned to participants who had not yet resumed normal activities by the end of the assessment period.
Time Frame: Day 1 through 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 524 | 515 | 196 | 201 | 217 | 193
days | 2.6 (3.8) | 2.0 (3.1) | 2.7 (4.1) | 2.1 (3.5) | 2.2 (3.2) | 2.5 (3.9)

29. Secondary Outcome: Mean Days Missed From Normal Activities in the Intent to Treat Population
Description: as for outcome 28
Time Frame: Day 1 through 14
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 585 | 584 | 234 | 238 | 236 | 230
days | 2.5 (3.7) | 2.1 (3.2) | 2.6 (4.0) | 2.1 (3.4) | 2.2 (3.2) | 2.7 (4.1)

30. Secondary Outcome: Number of Participants Reporting 1-14 Days of Analgesic Use in the Per Protocol Population
Description: As a quality of life measure, participants maintained a memory aid from Day 1 to Day 14 to track measures such as use of other, non-study medications such as analgesics. Each participant is summarized by the last day of reported analgesic usage, from the start of treatment with study intervention. The maximum number of days assessed, 14, was assigned to participants who were still taking analgesic medications by the end of the assessment period.
Time Frame: Day 1 through 14
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 533 | 524 | 198 | 203 | 218 | 193
participants
  Day 1 | 44 | 56 | 23 | 29 | 14 | 17
  Day 2 | 37 | 32 | 11 | 9 | 7 | 5
  Day 3 | 41 | 49 | 17 | 18 | 13 | 7
  Day 4 | 39 | 32 | 14 | 9 | 15 | 7
  Day 5 | 24 | 40 | 7 | 9 | 9 | 4
  Day 6 | 29 | 27 | 10 | 11 | 9 | 19
  Day 7 | 24 | 27 | 10 | 12 | 9 | 6
  Day 8 | 31 | 35 | 7 | 10 | 9 | 5
  Day 9 | 22 | 21 | 3 | 7 | 9 | 4
  Day 10 | 12 | 13 | 5 | 4 | 4 | 3
  Day 11 | 16 | 10 | 2 | 4 | 3 | 1
  Day 12 | 18 | 12 | 4 | 1 | 1 | 6
  Day 13 | 12 | 3 | 2 | 6 | 2 | 2
  Day 14 | 130 | 107 | 46 | 40 | 45 | 38

31. Secondary Outcome: Number of Participants Reporting 1-14 Days of Analgesic Use in the Intent to Treat Population
Description: as for outcome 30
Time Frame: Day 1 through 14
Population: All subjects who took at least one dose of study medication were included in the intent to treat population.
Measure: Number; unit: participants
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Number analyzed (Participants) | 617 | 630 | 250 | 249 | 248 | 248
participants
  Day 1 | 58 | 81 | 32 | 37 | 18 | 28
  Day 2 | 38 | 34 | 15 | 10 | 7 | 6
  Day 3 | 45 | 64 | 18 | 24 | 15 | 10
  Day 4 | 47 | 34 | 16 | 10 | 16 | 13
  Day 5 | 27 | 42 | 9 | 9 | 10 | 4
  Day 6 | 34 | 29 | 13 | 13 | 10 | 22
  Day 7 | 27 | 32 | 13 | 12 | 9 | 8
  Day 8 | 34 | 40 | 8 | 11 | 10 | 6
  Day 9 | 24 | 26 | 4 | 9 | 9 | 6
  Day 10 | 14 | 15 | 6 | 4 | 5 | 4
  Day 11 | 19 | 10 | 2 | 4 | 3 | 2
  Day 12 | 19 | 14 | 4 | 3 | 1 | 6
  Day 13 | 15 | 5 | 2 | 7 | 2 | 3
  Day 14 | 146 | 127 | 59 | 50 | 51 | 45

ADVERSE EVENTS:
Time Frame: All adverse events were recorded through the test of cure visit at Day 14-21; serious adverse events and new and recurrent skin infections were recorded though the extended follow-up visit at Day 49-63.
Arm/Group | Abscess, Placebo | Abscess, TMP/SMX | Infected Wound, TMP/SMX | Infected Wound, Clindamycin | Cellulitis, Cephalexin and TMP/SMX | Cellulitis, Cephalexin
Serious Adverse Events (participants affected / at risk) | 30/617 | 21/630 | 15/250 | 11/249 | 20/248 | 21/248
Other Adverse Events (participants affected / at risk) | 331/617 | 345/630 | 138/250 | 127/249 | 157/248 | 149/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abscess, Placebo (N=617) | Abscess, TMP/SMX (N=630) | Infected Wound, TMP/SMX (N=250) | Infected Wound, Clindamycin (N=249) | Cellulitis, Cephalexin and TMP/SMX (N=248) | Cellulitis, Cephalexin (N=248)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 8 (8) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Abscess limb (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 9 (9) | 5 (6) | 5 (5) | 1 (1) | 9 (10) | 11 (11)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coccidioidomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abscess, Placebo (N=617) | Abscess, TMP/SMX (N=630) | Infected Wound, TMP/SMX (N=250) | Infected Wound, Clindamycin (N=249) | Cellulitis, Cephalexin and TMP/SMX (N=248) | Cellulitis, Cephalexin (N=248)
Abdominal pain upper (Gastrointestinal disorders) | 26 (27) | 38 (40) | 17 (17) | 15 (20) | 19 (20) | 11 (11)
Abscess (Infections and infestations) | 130 (152) | 88 (100) | 20 (26) | 12 (13) | 27 (29) | 33 (39)
Cellulitis (Infections and infestations) | 5 (5) | 5 (5) | 6 (6) | 2 (2) | 27 (29) | 28 (28)
Constipation (Gastrointestinal disorders) | 16 (16) | 25 (25) | 17 (18) | 1 (1) | 7 (7) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 96 (102) | 94 (103) | 43 (48) | 81 (90) | 54 (59) | 47 (52)
Dizziness (Nervous system disorders) | 39 (41) | 41 (41) | 13 (14) | 13 (13) | 18 (20) | 16 (16)
Headache (Nervous system disorders) | 76 (81) | 100 (112) | 34 (36) | 27 (29) | 41 (45) | 42 (43)
Nausea (Gastrointestinal disorders) | 102 (112) | 134 (141) | 50 (56) | 28 (29) | 49 (51) | 41 (42)
Pyrexia (General disorders) | 25 (26) | 17 (17) | 2 (2) | 3 (3) | 13 (13) | 15 (16)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 16 (16) | 6 (6) | 4 (4) | 14 (14) | 5 (5)
Vomiting (Gastrointestinal disorders) | 40 (42) | 63 (64) | 22 (24) | 14 (14) | 19 (19) | 19 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less